CLINICAL TRIAL: NCT05914961
Title: ICK-Breast: Immunotherapy-related CRP Kinetics in Early and Metastatic Triple-negative Breast Cancer
Brief Title: Immunotherapy-related CRP Kinetics in Early and Metastatic Triple-negative Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Ulm (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Other Study IDs: ICK-Breast
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-04

CONDITIONS: TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample to assess laboratory parameters: Leukocytes, neutrophil granulocytes, lymphocytes, hemoglobin, hematocrit, thrombocytes, creatinin, glomerular filtration rate (GFR), serum glutamic oxaloacetic transaminase (GOT), serum glutamic pyruvic transaminase (GPT), bilirubin, lactate dehydrogenase (LDH), thyroid stimulating hormone (TSH), fT3 (free triiodothyronine), fT4 (free thyroxine), amylase, CRP, biomarkers related to immune response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Chemotherapy without immunotherapy
- Experimental Group: Chemotherapy in combination with immunotherapy

SUMMARY:
ICK-breast is a prospective, multicentric, non-interventional investigator-initiated trial (IIT) that aims to investigate the prognostic value of CRP kinetics in early and advanced or metastatic triple negative breast cancer (TNBC) under immune checkpoint inhibitor (ICI) therapy on pathological complete response (pCR) and event-free survival in early TNBC patients, and objective response rate (ORR), progression-free survival (PFS) and overall survival (OS) in advanced or metastatic TNBC.

DETAILED DESCRIPTION:
Immunotherapy, which involves activating the body's immune system for cancer treatment, has already been widely incorporated into the standard care of breast cancer patients with early and metastatic triple-negative breast cancer (TNBC).

This study aims to investigate how inflammatory markers such as C-reactive protein (CRP) change during and after immunotherapy. Study findings from other tumor types (kidney, lung, bladder) suggest that immunotherapy is particularly effective when a mild inflammatory response is triggered in the body. The investigators want to examine this using CRP measurement. CRP measurement can easily be integrated into clinical routine as it only requires a blood sample. And since the patients already need a blood draw for chemotherapy, CRP measurement can be performed directly from the blood sample.

The goal of this prospective study is to determine whether changes in CRP levels in the blood can predict the disease progression or response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* women ≥ 18 years of age
* histologically proven early or advanced or metastatic invasive breast cancer irrespective of therapy line
* ER-negative and progesterone receptor (PR)-negative and human epidermal growth factor receptor 2 (HER2)-negative (IHC 0-2+, Fluorescence In Situ Hybridization (FISH) neg.)
* patients with advanced or metastatic disease must be programmed cell death ligand 1 (PD-L1)-positive (IC ≥ 1 or combined positive score (CPS) ≥ 10) in the experimental group
* planned ICI therapy in combination with chemotherapy in the experimental group
* written informed consent into ICK-breast

Exclusion Criteria:

* ER-positive or PR-positive
* HER2-positive (IHC 2+, FISH pos or IHC 3+)
* any systemic breast cancer therapy before inclusion into the trial for early breast cancer patients
* any ICI therapy before inclusion into the trial
* pregnant or lactating patients
* inadequate general condition (not fit for chemotherapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 225 patients will be included in the study after written informed consent. Of 75 patients in the control group, which will undergo chemotherapy of physician's choice, 50 patients will be diagnosed with early TNBC and 25 patients will be diagnosed with advanced or metastatic TNBC.
  Of 150 patients in the experimental group, which will undergo chemotherapy in combination with ICIs, 100 patients will be diagnosed with early TNBC and 50 patients will be diagnosed with advanced or metastatic TNBC.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of CRP kinetics under ICI therapy on pathologic complete response (PCR) | duration of therapy and follow-up data (10 years)
  Evaluation of CRP kinetics to predict pCR in early (pathologic complete response) TNBC treated with ICI in combination with chemotherapy. The CRP value is determined from blood samples.

SECONDARY OUTCOMES:
Prognostic value of CRP kinetics under ICI therapy on objective response rate (ORR), progression free survival (PFS), event-free survival (EFS), invasive recurrence free survival and overall survival (OS) | duration of therapy and follow-up data (10 years)
  * evaluation of CRP kinetics to predict objective response in patients with metastatic TNBC receiving ICI in combination with chemotherapy
  * evaluation of CRP kinetics to predict progression free survival in patients with metastatic TNBC receiving ICI in combination with chemotherapy
  * evaluation of CRP kinetics to predict overall survival in patients with metastatic TNBC receiving ICI in combination with chemotherapy
  * evaluation of CRP kinetics to predict event-free survival in patients with early TNBC receiving ICI in combination with chemotherapy
  * evaluation of CRP kinetics to predict distant invasive recurrence free survival in patients with early TNBC receiving ICI in combination with chemotherapy The CRP value is determined from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Engler, Dr., Principal Investigator — Department of Women's Health Tübingen
Locations (1):
- Department of Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No